CLINICAL TRIAL: NCT04850300
Title: Efficiency Assessment of the Methodology for the Follow-up of Patients With Knee Prostheses
Acronym: PROknee
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Instituto de Investigacion Sanitaria INCLIVA (Other)
Responsible Party: Principal Investigator, Antonio Silvestre, Researcher and Head of the Orthopedic Surgery and Traumatology Service in Valencia University Clinical Hospital, Instituto de Investigacion Sanitaria INCLIVA
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020/181
Record Dates: First submitted 2021-04-08; First posted 2021-04-20 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Total Knee Arthroplasty
Keywords: Total knee arthroplasty; Functional assessment; Prognosis biomarkers; Medial condylar stabilization; Central pivot stabilization

STUDY DESIGN:
Intervention Model Description: This study describes a prospective triple-blinded, randomized, controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study participants, researchers who perform the functional assessments, and data analyst are unaware of the type of prosthetic stabilization used. They will not have access to the hospital medical history where the surgical procedure will be specified. The two surgeons in the study know the type of prosthesis used in each patient, and if the patient requests it, the technical specifications of the stabilization used are disclosed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total knee prosthesis 1 (Experimental): prosthesis with medial condylar stabilization
  Interventions: Procedure: Total knee prosthesis with medial condylar stabilization
- Total knee prosthesis 2 (Active Comparator): traditional prosthesis with central pivot stabilization
  Interventions: Procedure: Total knee prosthesis with central pivot stabilization

INTERVENTIONS:
Procedure: Total knee prosthesis with medial condylar stabilization — Surgery will be done of Total knee prosthesis with medial condylar stabilization
  Arms: Total knee prosthesis 1
Procedure: Total knee prosthesis with central pivot stabilization — Surgery will be done of Total knee prosthesis with central pivot stabilization
  Arms: Total knee prosthesis 2

SUMMARY:
Total knee arthroplasty (TKA) is currently the international standard for the treatment of degenerative and rheumatological diseases of the knee joint, as well as certain types of fractures. Although TKA is a procedure that has been shown to be effective in relieving pain and improving function in patients with osteoarthritis, approximately 20% of patients are dissatisfied with the results. Traditional methods of assessing the outcome after joint arthroplasty often focus on objective indicators of surgery and neglect the needs and opinions of patients. Because of this, this research project has the aim to know the effectiveness of two models of stabilization of total knee prostheses on the functionality achieved and perceived by the patient, as well as in the knee joint biomechanics during movement in activities of daily life. On the other hand, as a secondary objective, we propose to determine prognostic biomarkers of knee prosthesis function based on radiological information, quantification of cytokines, intra-articular markers, and biomechanical functional evaluation that correlate and predict a correct evolution of patients with a knee replacement.

To carry out these objectives, 80 participants will be included with an indication to perform total knee joint replacement surgery. Participants will be randomized allocated into two groups: i. participants with a prosthesis with medial condylar stabilization ii. participants with a traditional prosthesis with central pivot stabilization. Participants will be evaluated at five-times: before surgery, immediate postsurgical, at 3 months of evolution, 6 months of evolution, and one year of evolution.

DETAILED DESCRIPTION:
I. Objectives

Due to the information reviewed, this research project has the following aims:

1. To determine the effectiveness of two different prosthesis stabilization procedures of TKA on the functionality achieved and perceived by the patient, as well as on the knee joint biomechanics during movement in activities of daily life.
2. As a secondary objective, we propose to determine prognostic biomarkers of knee prosthesis function based on radiological information, quantification of cytokines, intra-articular markers, and biomechanical functional evaluation that correlate and predict a correct evolution of patients with knee replacements.

II. General procedures

The study has the approval of the Ethical Committee for Research with Drugs of the University Clinical Hospital of Valencia. Likewise, this study will be conducted at the University Clinical Hospital of Valencia with the INCLIVA Health Research Institute and the University of Valencia (Spain). All assessment procedures will be performed at the Evaluation Unit in Personal Autonomy, Dependence, and Mental Disorders of the Faculty of Medicine at the University of Valencia.

III. Methodology

III.1. Study design

The PROKnee trial was designed as a randomized, controlled, and triple-blinded (patient, raters, and data analysts) with two parallel groups.

III.2 Participants

The inclusion criteria are:

* People between 50-85 years old and,
* Primary total knee prosthesis surgery indication with patellar fitting.

The exclusion criteria are as follows:

* Previous lower limb joint prosthesis,
* History of fracture or surgery in the lower limb or lumbar spine,
* Disabling contralateral knee pain,
* Lower limb length asymmetry > 2 cm,
* Walking impairment due to other causes non-related to the knee pathology,
* Body Max Index > 39, and
* Severe surgical complications such as infection, aseptic loosening, deep vein thrombosis, periprosthetic fracture, and arthrofibrosis.

III.3 Assessment and Outcomes

The study participants will be evaluated in five periods of evolution: before surgery, immediately after surgery, at 3 months of evolution, at 6 months of evolution, and a year after having performed the surgery.

The set of tests to be carried out in each evaluation time and the data to be recorded are the following:

Personal and Anthropometric data:

* Age (years), Sex (men/women), Gender, BMI (kg/m2), race, level of education, marital status, height, weight, number of chronic diseases besides osteoarthritis, length of inferior extremities measured weight-bearing from the anterior iliac spine (AIS) to the medial malleolus, % of body fat, % of body water.
* Chronicity of knee symptoms; Diagnosis, Surgical approach, Prosthetic implant, Side of surgery, Days of hospital stay, Leg swelling evaluation with thigh and calf circumference, Hospital readmission, Post-cx complications, Fall Incidence.

Assessment scales:

* To assess knee and other joint pain it will be used the Visual Analog Scale (EVA).
* To assess knee function it will be used the Knee Osteoarthritis Outcome Score (KOOS).
* To assess pain, stiffness, and function it will be used the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).
* To assess physical activity it will be used the University of California, Los Angeles Physical Activity Questionnaire (UCLA).
* To assess health-related quality of life it will be used the EuroQol Group 5-dimensions-Level 5 (EQ5D5L) and the Short Form-12 Physical Functioning (SF-12).
* To assess cognitive state it will be used the Screen for Cognitive Impairment in Psychiatry (SCIP).
* To assess joint awareness it will be used the Forgotten joint score-12 (FJS-12).
* To assess anxiety and depression it will be used the Hospital Anxiety and Depression Scale (HADS).

Radiological and Laboratory tests:

* Imaging tests by radiography on the operated knee
* Carrying out computed tomography in cases of inadequate function, to identify possible causes, without subjecting the patients to excessive irradiation.
* Determination of Serum Levels of inflammatory biomarkers status: Interleukin-6, procalcitonin, calprotectin, and C-reactive protein.
* Determination of intra-joint biomarkers: C-reactive protein, and alpha-defensin.

Biomechanical functional assessment:

* Range of motion in both knees.
* Isometric knee strength flexion and extension of the operated and contralateral knee.
* Lower limb proprioception.
* Balance assessment during standing position.
* Kinematic assessment of the lower limb during 1) Six-minute walking test gait, 2) Timed up-and-go test, 3) Gait, 4) Sit to stand Test, 5) Step-over, 6) Stepping up and down stairs.

III.4 Intervention

Participants will be randomized and allocated into two groups: 1) participants with a prosthesis with medial condylar stabilization and, 2) participants with a traditional prosthesis with central pivot stabilization.

III.5 Sample size, recruitment, and randomization

The sample size was estimated based on previous works that compare the medial stabilization knee prosthesis with another device. A small-medium effect (f = 0.15), a statistical significance of 5% at the two-tailed level, and a power of 90% are set, which gives a total of 82 people to be recruited. If 20% of the possible dropouts are considered, the initial recruitment will be of 99 people. Because patient recruitment will occur over a prolonged period, the assignment to the groups will be performed as block randomization with a 1:1 allocation.

ELIGIBILITY:
The inclusion criteria are:

* People between 50-85 years old and,
* Primary total knee prosthesis surgery indication with patellar fitting.

The exclusion criteria are as follows:

* Previous lower limb joint prosthesis,
* History of fracture or surgery in the lower limb or lumbar spine,
* Disabling contralateral knee pain,
* Lower limb length asymmetry > 2 cm,
* Walking impairment due to other causes non-related to the knee pathology,
* Body Max Index > 39, and
* Severe surgical complications such as infection, aseptic loosening, deep vein thrombosis, periprosthetic fracture, and arthrofibrosis.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Maximum walking speed (MWS) | 1 year
  Maximum distance traveled by the body per unit of time (m·s-1). It will ask for participants to walk safely and as quickly as possible, without running, in a 10 m, straight and flat walkway. The two first and last stride will be discarded from the analysis in order to avoid the acceleration and deceleration of the star and end of the gait. The gait speed will be measured with the NedAMH/IBV v5.6 (Institute of Biomechanics of Valencia, Spain) software which uses two infrared or red light photocells to measured gait speed. This outcome will be measured in all the assessment times of the study.

SECONDARY OUTCOMES:
Self-reported pain | 1 year
  Measured with the Visual Analog Scale (EVA). High scores indicate higher pain sensations.
Self-reported knee function - Knee Osteoarthritis Outcome Score | 1 year
  Measured with the Knee Osteoarthritis Outcome Score (KOOS). It is a 42-item questionnaire, including 5 subscales: symptoms, pain, ADLs, sports/recreation, and quality of life. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Self-reported knee function - Western Ontario and McMaster Universities Osteoarthritis Index | 1 year
  Measured with the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). It is consisted of 33 items which evaluates the health and function of the patient from various aspects. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Higher scores are representative of better situation and less pain.
Self-reported Physical activity | 1 year
  Measured with the University of California, Los Angeles Physical Activity Questionnaire (UCLA). UCLA is a single-item 10-level-scale, ranging from level 10, representing a highly physically active patient, to level 1, a patient who is dependent on others and unable to leave home.
Joint awareness | 1 year
  Measured with the Forgotten joint score-12 (FJS-12) questionnaire; indicates the degree of discomfort that the patient perceives in the activities of daily living produced by the knee pathology. The FJS-12 contains 12 questions which are scored with a Likert scale ranging from 0 to 4. A lower score on the Likert scale equates to less awareness of the joint.
Health-related quality of life - EuroQol Group 5-dimensions-Level 5 | 1 year
  Measured with the EuroQol Group 5-dimensions-Level 5 (EQ5D5L). The test covers 5 dimensions of health (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with 5 levels of severity in each dimension (no problems, slight problems, moderate problems, severe problems, and unable to perform or extreme problems). Low scores on each item indicate a good perception of health.
Health-related quality of life - Short Form-12 Physical Functioning | 1 year
  Measured with the Short Form-12 Physical Functioning (SF-12). A higher score indicates higher levels of quality of life.
Mental status | 1 year
  Anxiety and depression will be measured with the Hospital Anxiety and Depression Scale (HADS). HADS is a fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression.
Cognitive status | 1 year
  Measured with the Screen for Cognitive Impairment in Psychiatry (SCIP) batery. High scores indicate better cognitive performance.
Range of motion | 1 year
  Active knee range of motion (º) and Passive knee range of motion (º) measured with a manual goniometer.
Muscle strength | 1 year
  Maximum muscle strength during knee flexion (N) and Maximum muscle strength during knee extension (N) registered with an electronic dynamometer.
Lowe limb proprioception | 1 year
  Measured by the number of degrees that the patient makes when equalizing a certain position with their legs. The more degrees of difference, the less proprioception the person being evaluated presents. Will be measured with the Physiological Profile Assessment tool.
Gait speed during the Six-minute walking test | 1 year
  Distance traveled by the body in six minutes (m·s-1).
Vertical range displacement of the Center of Masses during the Six-minute walking test | 1 year
  Range of vertical movement (displacement) performed by the center of mass during the test (mm).
Medial-lateral range displacement of the Center of Masses during the Six-minute walking test | 1 year
  Range of lateral movement (displacement) performed by the center of mass during the test (mm).
Medial-lateral Jerk during the Six-minute walking test | 1 year
  Lateral change rate of acceleration taken by the measured person while performing the test (m/s3)
Anterior-posterior Jerk during the Six-minute walking test | 1 year
  Anterior-posterior change rate of acceleration taken by the measured person while performing the test (m/s3)
Power Spectral Density in turning during the Six-minute walking test | 1 year
  Distribution of movement power over the frequency bands associated with movement during the trial (W/Hz).
Total execution time of Timed up and go test | 1 year
  Time spent by the person evaluated to perform the test (s)
Vertical range displacement of the Center of Masses during Timed up and go test | 1 year
  Range of vertical movement (displacement) performed by the center of mass during the test (mm).
Medial-lateral range displacement of the Center of Masses during Timed up and go test | 1 year
  Range of lateral movement (displacement) performed by the center of mass during the test (mm).
Medial-lateral Jerk during Timed up and go test | 1 year
  Lateral change rate of acceleration taken by the measured person while performing the test (m/s3)
Anterior-posterior Jerk during Timed up and go test | 1 year
  Anterior-posterior change rate of acceleration taken by the measured person while performing the test (m/s3)
Power Spectral Density in turning during Timed up and go test | 1 year
  Distribution of movement power over the frequency bands associated with movement during the trial (W/Hz).
Gait speed carried out in a 10-meter flat and unobstructed corridor | 1 year
  (ms-1)
Stride length during gait | 1 year
  Distance traveled by the person measured from the heel contact of one leg to the next heel contact of the same leg; measured in a 10-meter flat and unobstructed corridor with a 3D photogrammetry system and two dynamometric platforms (m).
Cadence during gait | 1 year
  Number of the steps calculated in a minute, measured in a 10-meter flat and unobstructed corridor with a 3D photogrammetry system and two dynamometric platforms (steps/min).
Stance time during gait | 1 year
  Percentage of the gait cycle that lasts the stance phase measured in a 10-meter flat and unobstructed corridor with a 3D photogrammetry system and two dynamometric platforms (% gait cycle).
Maximum knee extension during the stance phase of gait | 1 year
  Maximum knee extension achieved during the stance phase of gait measured in a 10-meter flat and unobstructed corridor with a 3D photogrammetry system (º).
Maximum knee flexion during the swing phase of gait | 1 year
  Maximum knee flexion achieved during the swing phase of gait measured in a 10-meter flat and unobstructed corridor with a 3D photogrammetry system (º).
Ground reaction force during weight acceptance of gait cycle | 1 year
  First peak of vertical force during stance phase of gait measured in a 10-meter flat and unobstructed corridor with a system of two dynamometric platforms (N).
Ground reaction force during toe-off of gait cycle | 1 year
  Second peak of vertical force during stance phase of gait measured in a 10-meter flat and unobstructed corridor with a system of two dynamometric platforms (N).
Maximum vertical force during Sit-to-stand test | 1 year
  Maximum vertical force of prosthetic leg and no-operated leg, calculated for sitting and standing phases separately; measured with a system of two dynamometric platforms (N).
Knee momentum during Sit-to-stand test | 1 year
  Product of knee mass and speed of movement performed for the prosthetic knee and no-operated knee, calculated for sitting and standing phases separately; measured with a 3D photogrammetry system (Nm).
Knee range of motion during Sit-to-stand test | 1 year
  Range of motion achieved by the prosthetic knee and no-operated knee, calculated for sitting and standing phases separately; measured with a 3D photogrammetry system (º).
Knee angular velocity during Sit-to-stand test | 1 year
  Rate of change of angular position with respect to time of the prosthetic knee and no-operated knee, calculated for sitting and standing phases separately; measured with a 3D photogrammetry system (º/seg).
Maximum vertical ground reaction force in the single stance of the Step-over test | 1 year
  Maximum vertical ground reaction force in the single stance over the step for the prosthetic and no-operated knee, measured with a system of two dynamometric platforms (N)
Maximum vertical ground reaction force in landing phase of the Step-over test | 1 year
  Maximum vertical ground reaction force in landing for the prosthetic and no-operated knee, measured with a system of two dynamometric platforms (N)
Knee momentum during the single stance phase of the Step-over test | 1 year
  Product of knee mass and speed of movement performed during the single stance step for the prosthetic and no-operated knee, measured with a 3D photogrammetry system (Nm)
Knee range of motion Step-over test | 1 year
  Range of motion achieved during the trial for the prosthetic and no-operated knee, measured with a 3D photogrammetry system (º)
Knee angular velocity during swing phase of the Step-over test | 1 year
  Rate of change of angular position with respect to time for the prosthetic and no-operated knee, during the swing phase of step over, measured with a 3D photogrammetry system (º/s)
Maximum knee flexion from Stepping up and down stairs test | 1 year
  Maximum knee flexion during up and down for the prosthetic and no-operated knee and measured with a 3D photogrammetry system (º)
Knee angular velocity from Stepping up and down stairs test | 1 year
  Rate of change of angular position with respect to time during up and down, for the prosthetic and no-operated knee and measured with a 3D photogrammetry system (º/s)
Maximum vertical ground reaction force in single support from Stepping up and down stairs test | 1 year
  Maximum vertical ground reaction force in single support during up and down for the prosthetic and no-operated knee and measured with two dynamometric platforms (N).
Flexion/extension knee momentum in up and down from Stepping up and down stairs test | 1 year
  Product of knee mass and speed of movement performed for the prosthetic and no-operated knee and measured with a 3D photogrammetry system (Nm).
Varus/valgus knee momentum during up and down from Stepping up and down stairs test | 1 year
  Product of knee mass and speed of movement performed for the prosthetic and no-operated knee and measured with a 3D photogrammetry system (Nm).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Silvestre Muñoz, PhD., Principal Investigator — Orthopedic Surgery and Traumatology Service of the University Clinical Hospital of Valencia, Spain.
Locations (2):
- Spain (2):
  - Orthopedic Surgery and Traumatology Service of the University Clinical Hospital of Valencia, Valencia
  - Unidad de Evaluación en Autonomía Personal, Dependencia y Trastornos Mentales Graves (TMAP), University of Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poley González A, Ortega Blanco JA, Pedregal González M, Martín Azofra M, Hermosilla Camacho C, Mora Moreno F. Prevalencia de enfermedades osteoarticulares y consumo de recursos. Calidad de vida y dependencia en pacientes con artrosis. Med Fam SEMERGEN. 2011;37(9):462-7.
- [Background] Rodríguez-Merchán EC, Oussedik S, editores. Total Knee Arthroplasty: A Comprehensive Guide. Springer International Publishing; 2015.
- [Background] Maradit Kremers H, Visscher SL, Moriarty JP, Reinalda MS, Kremers WK, Naessens JM, Lewallen DG. Determinants of direct medical costs in primary and revision total knee arthroplasty. Clin Orthop Relat Res. 2013 Jan;471(1):206-14. doi: 10.1007/s11999-012-2508-z. PMID 22864619
- [Background] Coles T, Williams V, Dwyer K, Mordin M. Psychometric Evaluation of the Patient's Knee Implant Performance Questionnaire. Value Health. 2018 Nov;21(11):1305-1312. doi: 10.1016/j.jval.2018.05.006. Epub 2018 Jun 30. PMID 30442278
- [Background] Behrend H, Giesinger K, Giesinger JM, Kuster MS. The "forgotten joint" as the ultimate goal in joint arthroplasty: validation of a new patient-reported outcome measure. J Arthroplasty. 2012 Mar;27(3):430-436.e1. doi: 10.1016/j.arth.2011.06.035. Epub 2011 Oct 13. PMID 22000572
- [Background] Rousseau MA, Lazennec JY, Catonne Y. Early mechanical failure in total knee arthroplasty. Int Orthop. 2008 Feb;32(1):53-6. doi: 10.1007/s00264-006-0276-7. Epub 2006 Nov 21. PMID 17119961
- [Background] Ito H, Ichihara K, Tamari K, Amano T, Tanaka S, Uchida S. Factors characterizing gait performance of patients before and soon after knee arthroplasty. J Phys Ther Sci. 2021 Mar;33(3):274-282. doi: 10.1589/jpts.33.274. Epub 2021 Mar 17. PMID 33814716
- [Background] Ro DH, Han HS, Lee DY, Kim SH, Kwak YH, Lee MC. Slow gait speed after bilateral total knee arthroplasty is associated with suboptimal improvement of knee biomechanics. Knee Surg Sports Traumatol Arthrosc. 2018 Jun;26(6):1671-1680. doi: 10.1007/s00167-017-4682-8. Epub 2017 Aug 28. PMID 28849392
- [Background] Rosello Anon A, Martinez Garrido I, Cervera Deval J, Herrero Mediavilla D, Sanchez Gonzalez M, Vicent Carsi V. Total ankle replacement in patients with end-stage ankle osteoarthritis: clinical results and kinetic gait analysis. Foot Ankle Surg. 2014 Sep;20(3):195-200. doi: 10.1016/j.fas.2014.04.002. Epub 2014 Apr 18. PMID 25103708
- [Derived] San Martin Valenzuela C, Tabares-Seisdedos R, Paya Rubio A, Correa-Ghisays P, Pedrero-Sanchez JF, Silvestre Munoz A. Efficiency assessment of follow-up methodology of patients with knee replacement to predict post-surgical functionality: a protocol for randomised control PROKnee trial. BMJ Open. 2024 May 7;14(5):e077942. doi: 10.1136/bmjopen-2023-077942. PMID 38719321